CLINICAL TRIAL: NCT00290615
Title: Phase II Study of Oxaliplatin, Capecitabine, Cetuximab, and Bevacizumab in the Treatment of Metastatic Colorectal Cancer
Brief Title: Capecitabine, Cetuximab, Oxaliplatin, and Bevacizumab in Treating Patients With Metastatic or Recurrent Colorectal Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Hurwitz (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007431 (CDR0000449945); DUMC-7118-05-4R0
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; recurrent colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Cetuximab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine, Oxaliplatin, Bevacizumab, Cetuximab (Experimental): Capecitabine - oral administration of 850 mg/m2 every 12 hours on days 1-14. Oxaliplatin - IV administration of 130 mg/m2 over 2 hours on day 1 of a cycle. Bevacizumab- IV administration of 7.5 mg/kg over 30-90 minutes on day 1 of a cycle.
  Cetuximab at an initial dose of 400 mg/m2 over 120 minutes and subsequently 250 mg/m2 over 60 minutes on day 1 of a cycle.
  Cycles are 21 days.
  Interventions: Biological: bevacizumab; Biological: cetuximab; Drug: capecitabine; Drug: oxaliplatin

INTERVENTIONS:
Biological: bevacizumab
  Other Names: Avastin
Biological: cetuximab
Drug: capecitabine
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as cetuximab and bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab and bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving capecitabine together with cetuximab, oxaliplatin, and bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving capecitabine together with cetuximab, oxaliplatin, and bevacizumab works in treating patients with metastatic or recurrent colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with unresectable metastatic or recurrent colorectal adenocarcinoma treated with capecitabine, cetuximab, oxaliplatin, and bevacizumab.

Secondary

* Determine the safety and tolerability of this regimen in these patients.
* Determine the progression-free and overall survival of patients treated with this regimen.

Exploratory

* Determine the effect of this regimen on the angiogenesis biomarkers in these patients.
* Determine the effect of this regimen on wound angiogenesis in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral capecitabine twice daily on days 1-14. Patients will also receive cetuximab IV over 1-2 hours, oxaliplatin IV over 2 hours, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 1 month.

PROJECTED ACCRUAL: Approximately 45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Unresectable disease
  * Metastatic or recurrent disease
* Not amenable to potentially curative treatment
* No untreated leptomeningeal or brain metastases

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* No known uncontrolled coagulopathy

Hepatic

* AST and ALT < 2.5 times upper limits of normal (ULN) (5 times ULN if liver metastases are present)
* Bilirubin < 2.0 times ULN

Renal

* Creatinine clearance > 40 mL/min
* Urine protein negative
* Urine protein:creatinine ratio > 1

Cardiovascular

* No unstable or uncontrolled hypertension (i.e., blood pressure [BP] > 150/100 mm Hg despite antihypertensive therapy)

  * Patients who recently started or have adjusted antihypertensive medications are eligible provided BP is < 140/90 mm Hg for ≥ 3 different measurements over 14 days
* No arterial thromboembolic events within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction
  * Clinically significant peripheral vascular disease
* No New York Heart Association class III-IV congestive heart failure
* No uncontrolled symptomatic coronary artery disease or cardiac arrhythmia
* No other significant uncontrolled cardiac disease

Gastrointestinal

* No lack of physical integrity of the upper gastrointestinal tract
* No malabsorption syndrome
* No inability to tolerate oral medication

Immunologic

* No prior severe infusion reaction to a monoclonal antibody
* No history of an allergic reaction attributed to compounds of similar chemical or biologic composition to oxaliplatin, cetuximab, capecitabine, or bevacizumab
* No prior unanticipated, severe reaction to fluoropyrimidine therapy or known hypersensitivity to fluoroucacil

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during the study and for 3-4 months after completion of study treatment
* No peripheral neuropathy ≥ grade 2
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No known dihydropyrimidine dehydrogenase deficiency

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior adjuvant bevacizumab or cetuximab
* No other concurrent anticancer immunotherapy or biologic therapy

Chemotherapy

* At least 6 months since a prior adjuvant fluorouracil-, leucovorin calcium-, or capecitabine-based regimen
* At least 12 months since prior adjuvant oxaliplatin
* No prior chemotherapy for metastatic or recurrent disease

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery and recovered
* More than 6 months since vascular surgery, stenting, or angioplasty

Other

* At least 4 weeks since prior and no concurrent sorivudine or brivudine
* More than 4 weeks since prior participation in any investigational drug study
* No prior therapy that affects or targets the epidermal growth factor pathway
* No concurrent cimetidine

  * Concurrent ranitidine, famotidine, or proton-pump inhibitors allowed
* Concurrent anticoagulation therapy with full-dose anticoagulant allowed provided dose is stable for at least 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I. Hurwitz, MD, Study Chair — Duke Cancer Institute
Locations (2):
- United States (2):
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina

REFERENCES:
- [Result] Wong NS, Fernando NH, Nixon AB, Cushman S, Aklilu M, Bendell JC, Morse MA, Blobe GC, Ashton J, Pang H, Hurwitz HI. A phase II study of capecitabine, oxaliplatin, bevacizumab and cetuximab in the treatment of metastatic colorectal cancer. Anticancer Res. 2011 Jan;31(1):255-61. PMID 21273607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between October 2005 and June 2007 in the Duke Cancer Center, Duke Oncology Network, and Wake Forest University.
Period: Overall Study
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab, Cetuximab
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab, Cetuximab
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Percentage of Participants With Partial or Complete Response)
Description: Restaging scans occurred every 9 weeks from time of study drug initiation until disease progression.
  Disease assessment was performed and recorded according to the Response Evaluation Criteria in Solid Tumors (RECIST v.1.0) Guidelines.
  The definitions were:
  Complete response (CR)- Disappearance of all target lesions Partial response (PD)- At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Stable disease (SD)- Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started Progressive disease (PD) - At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: After all subjects were evaluated for restaging which occured every 9 weeks from drug initiation until disease progression, assesed up to 24 months.
Population: All subjects who received restaging scans were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab, Cetuximab
Number analyzed (Participants) | 30
percentage of participants with response | 43 [25 to 63]

2. Secondary Outcome: Safety and Tolerability
Description: Number of participants with adverse events
Time Frame: After all participants went off study drug regimine.
Measure: Number; unit: participants with adverse event
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab, Cetuximab
Number analyzed (Participants) | 30
participants with adverse event | 30

3. Secondary Outcome: Progression-free Survival
Description: Disease assessment was performed and recorded according to the Response Evaluation Criteria in Solid Tumors (RECIST v.1.0) Guidelines.
  Progressive disease is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  This is the average number of months participants survived without showing progressive disease.
Time Frame: From time of treatment until documented progression or death from any cause, whichever came first, assesed up to 60 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab, Cetuximab
Number analyzed (Participants) | 30
months | 10.3 [6.8 to 16.3]

4. Other Pre Specified Outcome: Effect on Angiogenesis Biomarkers
Time Frame: After study completion
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Effect on Wound Angiogenesis
Time Frame: After study completion
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival
Description: Average months of survival of participants after receiving study drug.
Time Frame: From time of treatment until death from any cause, assesed up to 60 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab, Cetuximab
Number analyzed (Participants) | 30
months | 18.8 [14.2 to 23.7]

ADVERSE EVENTS:
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab, Cetuximab
Serious Adverse Events (participants affected / at risk) | 10/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine, Oxaliplatin, Bevacizumab, Cetuximab (N=30)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated ALT/AST (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 2 (2)
Bowel obstruction (Gastrointestinal disorders) | 2 (2)
Bowel perforation (Gastrointestinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep Venous Thrombosis (Vascular disorders) | 1 (1)
Death (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine, Oxaliplatin, Bevacizumab, Cetuximab (N=30)
Neutropenia (Blood and lymphatic system disorders) | 10 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (15)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Thromboembolism (Vascular disorders) | 4 (4)
Skin rash (Skin and subcutaneous tissue disorders) | 27 (27)
Sensory neuropathy (Nervous system disorders) | 25 (25)
Proteinuria (Renal and urinary disorders) | 6 (6)
Paronychia (Skin and subcutaneous tissue disorders) | 3 (3)
Hypomagnesium (Metabolism and nutrition disorders) | 17 (17)
Hypertension (Vascular disorders) | 3 (3)
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 7 (7)
Fatigue (General disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 15 (15)
Diarrhea (Gastrointestinal disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No